CLINICAL TRIAL: NCT06463990
Title: Association Between the Triglyceride-glucose Index and the Ratio of Triglyceride to High-density Lipoprotein Cholesterol With Fetal Macrosomia in Low-risk Nulliparous Pregnant Women
Brief Title: Influence of TyG Index and TG/HDL-C Ratio on Fetal Macrosomia
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Fahri Burcin Firatligil, Specialist doctor in obstetrics and gynecology and Fellow student in Perinatology, Ankara Etlik City Hospital
Other Study IDs: AECH-FIRATLIGIL-001
Record Dates: First submitted 2024-06-08; First posted 2024-06-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Fetal Macrosomatia; Lipid Metabolism Disorders; Hyperlipidemias
Keywords: Fetal macrosomia; Nulliparous; Triglyceride; TyG index
MeSH Terms: conditions — Lipid Metabolism Disorders; Hyperlipidemias; Fetal Macrosomia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Singleton nulliparous pregnant women who had performed an oral glucose challenge test (OGCT) between 24 and 28 weeks' gestation with a result of less than 140 mg/dL had blood samples taken at 8:00 am on the first visit to the outpatient clinic in the third trimester after an 8-hour fasting state
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: women with macrosomic newborns
  Interventions: Other: TyG index
- Control group: women with non-macrosomic newborns
  Interventions: Other: TyG index

INTERVENTIONS:
Other: TyG index — association between TyG index and triglyceride to high-density lipoprotein cholesterol ratio with fetal macrosomia
  Other Names: Triglyceride to high-density lipoprotein cholesterol ratio

SUMMARY:
Metabolic disorders that can occur during pregnancy, in particular disorders of lipid metabolism and insulin resistance, can have a detrimental effect on pregnancy and the fetus.

The triglyceride level and other lipids increase slightly during pregnancy. This increase has a positive effect on the development of the fetus. However, an excessive increase in lipid levels can cause some metabolic disorders such as gestational diabetes and increase feto-maternal morbidity/mortality.

While some existing studies have shown that elevated triglyceride levels can cause fetal macrosomia, others have found no correlation between these two variables. The ratio of triglycerides to HDL is a widely used marker for lipid disorders. In addition, the triglyceride-glucose index is also an index used to detect insulin resistance.

DETAILED DESCRIPTION:
In this study, the investigators aimed to investigate whether the ratio of triglycerides to high-density lipoprotein cholesterol and the triglyceride glucose index are associated with fetal macrosomia in low-risk nulliparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Screening for fetal macrosomia was based on the term defined according to the standards of the American College of Obstetricians and Gynecologists (ACOG).
* Low-risk nulliparous singleton pregnant women.
* Age between 18 and 40 years old

Exclusion Criteria:

* Post-term pregnancies
* Hospitalized for preterm labor or preterm premature rupture of membranes.
* Gestational diabetes mellitus, diabetes mellitus type I - type II.
* Pregnant women with fetal growth restriction, hypertensive pregnancy disorders, familial hypercholesterolemia and hyperlipidemia.
* Multiparous pregnant women
* Multiple pregnancies
* Pregnant women with chronic diseases.
* Pregnant women with impaired liver function;
* Pregnant women with body mass index <25 and >40 kg/m2.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The singleton pregnant women who delivered a macrosomic newborn were included in the study group (Group I) and the singleton pregnant women who delivered a non-macrosomic fetus were included in the control group (Group II). For each pregnant woman who met the inclusion and exclusion criteria and was eligible for Group I, the first patient in the ranking order of the files who met the criteria previously mentioned in the Materials and Methods section was selected for Group II.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
The TyG index | between 28 and 40 weeks of pregnancy
  The triglyceride-glucose index was determined using the formula Ln [fasting triglycerides (mg/dL) × fasting plasma glucose (mg (dL)/2], with blood samples taken from pregnant women in the third trimester.
The triglyceride to high density lipoprotein cholesterol ratio | between 28 and 40 weeks of pregnancy
  The triglyceride to high density lipoprotein cholesterol ratio was calculated from the blood samples taken from pregnant women in the third trimester.

SECONDARY OUTCOMES:
HOMA-IR | between 28 and 40 weeks of pregnancy
  HOMA-IR was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5 with blood samples taken from pregnant women in the third trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Yaprak Engin-Ustun, Prof, Study Director — Etlik Zubeyde Hanim Women's Health Education and Research Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data are available on request only due to ethical, legal or commercial reasons
Supporting Information: Analytic Code
Time Frame: one or two months

REFERENCES:
- [Result] Macrosomia: ACOG Practice Bulletin, Number 216. Obstet Gynecol. 2020 Jan;135(1):e18-e35. doi: 10.1097/AOG.0000000000003606. PMID 31856124
- [Result] Poveda NE, Garces MF, Darghan AE, Jaimes SAB, Sanchez EP, Diaz-Cruz LA, Garzon-Olivares CD, Parra-Pineda MO, Bautista-Charry AA, Muller EA, Alzate HFS, Acosta LMM, Sanchez E, Ruiz-Parra AI, Caminos JE. Triglycerides/Glucose and Triglyceride/High-Density Lipoprotein Cholesterol Indices in Normal and Preeclamptic Pregnancies: A Longitudinal Study. Int J Endocrinol. 2018 Aug 6;2018:8956404. doi: 10.1155/2018/8956404. eCollection 2018. PMID 30158976
- [Result] Babic N, Valjevac A, Zaciragic A, Avdagic N, Zukic S, Hasic S. The Triglyceride/HDL Ratio and Triglyceride Glucose Index as Predictors of Glycemic Control in Patients with Diabetes Mellitus Type 2. Med Arch. 2019 Jun;73(3):163-168. doi: 10.5455/medarh.2019.73.163-168. PMID 31404127
- [Result] Barat S, Ghanbarpour A, Bouzari Z, Batebi Z. Triglyceride to HDL cholesterol ratio and risk for gestational diabetes and birth of a large-for-gestational-age newborn. Caspian J Intern Med. 2018 Fall;9(4):368-375. doi: 10.22088/cjim.9.4.368. PMID 30510652
- [Derived] Firatligil FB, Tuncdemir S, Sucu S, Reis YA, Ozkan S, Dereli ML, Sucu ST, Engin-Ustun Y. Association of the triglyceride-glucose index and the ratio of triglyceride to high-density lipoprotein cholesterol with fetal macrosomia in nulliparous pregnant women: a prospective case-control study. BMC Pregnancy Childbirth. 2025 Feb 17;25(1):175. doi: 10.1186/s12884-025-07317-5. PMID 39962459